CLINICAL TRIAL: NCT03555786
Title: Minimum Effective Volume of Bupivacaine for Retroclavicular Approach Brachial Plexus Block
Brief Title: MEV for Retroclavicular Approach to Infraclavicular Block
Status: Terminated | Type: Observational
Why Stopped: Failure of recruitment
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AntalyaTRH25
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2018-11

CONDITIONS: Bupivacaine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: minimum effective volume — The determination of MEV90 and its 95% confidence interval (CI) will be based on a "biased coin up-and-down sequential design

SUMMARY:
In this study, the primary objective was to estimate the minimum effective volume of bupivacaine 0.5% resulting in successful block in 90% of patients (MEV90) for ultrasound-guided retroclavicular approach to infraclavicular brachial plexus block.

DETAILED DESCRIPTION:
A "biased coin up-and-down sequential design" will be applied to assess the minimum effective volume in 90% of patients for the retroclavicular brachial plexus block. The first subject received 25 ml 0.5% bupivacaine . Each subsequent patient received a dose that depended on the response of the previous one. If the previous block is successful, the block will be performed either by a reduction of the volume by 2.5 ml with a probability ß = 0.11 or by a same dose of the previous one with a probability 1-ß = 0.89 in the next patient.

ELIGIBILITY:
Inclusion Criteria:

* patients who received infraclavicular brachial plexus block for elective elbow, forearm, wrist, or hand surgery
* American Society of Anesthesiologists class I, II or III

Exclusion Criteria:

* patients <18 years old
* >65 years old
* body mass index (BMI) <20 or >35 kg/m2
* inability to provide written informed consent
* refusal of regional anesthesia
* pregnancy
* contraindication for regional anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between 18 and 65 years of age with infraclavicular brachial lexus block for elective elbow, forearm, wrist, or hand surgery , were selected in the study.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
The minimum effective volume of bupivacaine 0.5% resulting in successful block in 90% of patients (MEV90) | 30 minutes
  The determination of MEV90 and its 95% confidence interval (CI) will be based on a "biased coin up-and-down sequential design

CONTACTS AND LOCATIONS:
Overall Officials: Ali Sait Kavakli, MD, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)